CLINICAL TRIAL: NCT00720590
Title: Effect of HIV-1 Protease Inhibitors on Endothelial Function and Glucose Metabolism in Normal, HIV-Uninfected Subjects: Atazanavir or Lopinavir/Ritonavir or Placebo
Brief Title: Effect of the HIV Protease Inhibitors Atazanavir and Lopinavir/Ritonavir on Cardiovascular Disease Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Michael P. Dubé, MD, Indiana University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 573; R01HL072711 (NIH); R01HL072711-01 (NIH)
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2008-07

CONDITIONS: Endothelial Dysfunction
MeSH Terms: interventions — Atazanavir Sulfate; Lopinavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants will receive treatment with atazanavir and placebo lopinavir/ritonavir.
  Interventions: Drug: Atazanavir; Drug: Placebo
- 2 (Experimental): Participants will receive treatment with lopinavir/ritonavir and placebo atazanavir.
  Interventions: Drug: Lopinavir/ritonavir; Drug: Placebo
- 3 (Placebo Comparator): Participants will receive treatment with placebos for both drugs.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atazanavir — 400 mg of atazanavir (two 200-mg capsules) per day for 4 weeks
  Arms: 1
Drug: Lopinavir/ritonavir — 400 mg/100 mg of lopinavir/ritonavir (three soft-gel capsules, each containing 133.3 mg lopinavir and 33.3 mg ritonavir) twice per day with food for 4 weeks
  Arms: 2
Drug: Placebo — Daily dose of placebo for 4 weeks

SUMMARY:
HIV protease inhibitors (PIs) are a class of antiretroviral drugs used to inhibit viral replication. They do so by interfering with a key step in the replication process. Some HIV PIs have been associated with an increased risk of adverse cardiovascular side effects. Further study is needed, however, to assess the full extent of effect of newer HIV PIs, including atazanavir and lopinavir/ritonavir, on cardiovascular disease risk. This study will compare the effects of atazanavir, lopinavir/ritonavir, and placebo on certain cardiovascular disease risk factors in healthy people without HIV.

DETAILED DESCRIPTION:
Antiretroviral therapy for HIV, particularly with the use of PIs, is associated with an increased risk of heart attack. Specific cardiovascular side effects seen with the use of some PIs include insulin resistance, abnormal blood lipid levels, and endothelial dysfunction (abnormalities in the cells that line the inner surface of blood vessels). Past studies have shown that treatment with indinavir, an older PI, results in significant endothelial dysfunction, which may be the main cause for the increase in cardiovascular risk. Indinavir is now seldom used in clinical practice, and the newer PIs atazanavir and combination lopinavir/ritonavir now account for nearly 70% of total PI use in the United States. It is not known what effect these new PIs have on endothelial dysfunction. This study will compare the effects of atazanavir, lopinavir/ritonavir, and placebo on certain cardiovascular disease risk factors, including abnormal glucose metabolism and endothelial dysfunction, in healthy people without HIV.

Participation in this study will last 4 weeks. All participants will undergo initial assessments that will include various vascular and metabolic evaluations. Body weight, height, basal heart rate, and systolic and diastolic blood pressure will also be measured. Participants will then be assigned randomly to receive 4 weeks of treatment with 400 mg of atazanavir per day plus placebo, 400 mg/100 mg of lopinavir/ritonavir twice per day plus placebo, or placebos for both drugs per day. Upon completing the 4 weeks of treatment, participants will repeat the initial assessments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and lean with normal lipids
* Not infected with HIV or viral hepatitis

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-11; Primary Completion 2006-09 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Leg blood flow response to the intra-femoral artery infusion of methacholine chloride | Measured at Week 4

SECONDARY OUTCOMES:
Insulin sensitivity measured by the hyperinsulinemic euglycemic clamp study | Measured at Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Dubé, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Dube MP, Shen C, Greenwald M, Mather KJ. No impairment of endothelial function or insulin sensitivity with 4 weeks of the HIV protease inhibitors atazanavir or lopinavir-ritonavir in healthy subjects without HIV infection: a placebo-controlled trial. Clin Infect Dis. 2008 Aug 15;47(4):567-74. doi: 10.1086/590154. PMID 18636958